CLINICAL TRIAL: NCT05115929
Title: Standard Craniectomy Against Laparotomy for the Treatment of Traumatic Rise in Intracranial Pressure and the Effect on Long-term Outcome
Acronym: SCALPEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Federal Ministry of Defence (Germany) (Unknown); Bundesministerium der Verteidigung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021_10_SK1
Record Dates: First submitted 2021-10-10; First posted 2021-11-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Traumatic Brain Injuries
Keywords: Traumatic Brain Injuries; Decompressive Craniectomy; Decompressive Laparotomy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Decompressive Craniectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive Craniectomy Group (Active Comparator): participants with severe TBI randomly assigned as described in the study protocol
  Interventions: Procedure: Decompressive Craniectomy
- Decompressive Laparotomy Group (Active Comparator): participants with severe TBI randomly assigned as described in the study protocol
  Interventions: Procedure: Decompressive Laparotomy

INTERVENTIONS:
Procedure: Decompressive Laparotomy — As described in the study protocol a long midline laparotomy is performed and open abdomen therapy using negative pressure dressings initiated to lower abdominal pressure and thereby improve venous return from the brain to lower intracranial pressure.
  Arms: Decompressive Laparotomy Group
Procedure: Decompressive Craniectomy — As described in the study protocol a sufficiently sized hemi-craniectomy is performed and the skin closed over the bony defect to allow cerebral swelling and thereby lower intracranial pressure.
  Arms: Decompressive Craniectomy Group

SUMMARY:
Intractable high intracranial pressures (ICP) are associated with poor functional outcomes and mortality, so the SCALPEL trials aims to evaluate the effect of decompressive craniectomy against decompressive laparotomy to lower those pressures in diffuse TBI. The primary outcome measure for that evaluation is functional outcome after 12 months on the extended Glasgow Outcome Scale (GOS-E).

DETAILED DESCRIPTION:
Rationale for trial:

Traumatic brain injuries (TBI) are held responsible for about half of the trauma related death rate and a main driver of trauma related morbidity. While outcomes from trauma have improved in the last decades, the mortality and morbidity caused by TBI stayed about the same.

The surgical interventions for raised ICP in TBI have been studied extensively with varying outcome. Craniectomy did reduce mortality in several trials. There were additional survivors with favorable neurological outcome, as well as additional survivors with poor functional outcome. That effect might partly be explained by the inherent morbidity of the craniectomy or the consecutive cranioplasty. Various studies have shown surgical complications post cranioplasty in around one third of the cases including reoperation for hematoma, hydrocephalus, seizures, and graft infections and there is evidence for negative effects due to the rapid decompression of the pressure as growing hematoma size.

Decompressive laparotomy (DL) on the other side is thought to lower not only the dynamic pulsatile effect on the brain, it also causes increased venous outflow from the brain which reduces the intracranially present amount of venous blood and therefore ICP.

It is hypothesized that a decompressive laparotomy may have the benefit of lowering the ICP, without the inherent risks and complications caused by a large craniectomy and its influence on long-term outcome.

This trial seeks to inform future guidelines about this potentially alternative intervention in TBI patients. Another potential benefit might be in the applicability of the findings in settings without neurosurgical capabilities (expertise or instruments) like in military conflicts, rural areas, or developing countries.

If the treating team involving a neurosurgeon and a general, abdominal, or trauma surgeon depending on the local setting and jurisdiction agree that the participant matches the eligibility criteria, consent is given and no exclusion criteria are met, the participant can be enrolled in the trial.

Enrolment of a participant:

If a potential participant is admitted to a study center the local principal investigator (PI) is informed. If the local team is uncertain about eligibility or exclusion, advice from a senior clinician of the trial management committee (TMC) will be provided.

If after all there is still uncertainty about the potential eligibility, the patient will not be enrolled in the trial.

By definition the included participants will be unable to give written consent to participation in this study. In those cases, the investigators plan to discuss the procedures and the trial with the next of kin and acquire consent for the participant.

There are cases imaginable when the next of kin is unknown, cannot be reached, or there is no time to arrive and have that detailed discussion, due to the emergence of that immediate life-threatening condition. Those situations are covered by the Declaration of Helsinki. Detailed standard operating procedures as discussed in the SCALPEL Study Protocol, will be put in place together with the participating centers and the ethical monitoring board.

The investigators plan to set up 10 international centers in order to increase external validity of the trial and to complete the inclusion phase within 3 years.

Study Intervention:

The medical and interventional therapies included in step I and II are representing the current standard of care and are discussed extensively in the guidelines for severe traumatic brain injuries.

Step I includes head elevation 30-45°, adequate sedation, neuroprotective ventilation, sufficient analgesia and the use of vasopressors if necessary to support cerebral perfusion pressure. Monitoring includes measurement of ICP, IAP, and mean airway pressure. Those measures are all considered to be mandatory before progressing to randomization.

Step II includes ventriculostomy and drainage of CSF, infusion of mannitol or hypertonic saline, as well as therapeutic hypothermia. Those measures are considered to be facultative. The latter two are not of proven value, or might even be harmful, so the local team can very well skip those measures with respect to the local centers guidelines.

If the ICP remains over 25 mmHg for 1-12h and the inclusion criteria are met, without any exclusion criteria the patient can be randomized in the surgical intervention groups.

If randomized to the craniectomy treatment arm, it is discretionary to the treating neurosurgeon if a bifrontal vs. frontotemporoparietal hemicraniectomy is performed, depending on the clinical situation and local protocols. The bone flap should be generous. Secondary to the decompression there will be the necessity for a cranioplasty after resolving of the brain swelling 2 to 20 weeks after craniectomy.

The performance of the decompressive craniectomy is described in the Appendix B of the SCALPEL Study Protocol - Best practice guideline for the decompressive craniectomy in the SCALPEL trial.

If randomized to the laparotomy treatment arm, A long median laparotomy will be performed in the laparotomy group. The skin and fascia is left open after that as a laparostomy. It is covered by a negative pressure dressing or other adequate laparostomy dressings according to the local protocols. A traction-free mesh should be used with the fascial edges.

To further improve the procedural safety and effectiveness the investigators plan to monitor the effect on ICP for one hour directly in the operating theater after the negative pressure dressing is applied and before the patient is transferred to the neurosurgical ICU. Neurocritical care measures like head elevation 30-45°, adequate sedation, neuroprotective ventilation, sufficient analgesia and the use of vasopressors if necessary to support cerebral perfusion pressure, will be performed during that period as it would be done on the ICU ward.

Secondary to the decompression the closure of the fascia and skin is needed. If the ICP and neurological recovery of the patient allows, it is encouraged to perform the closure around 7-14 days after decompression. In the case-control study out of the Shock Trauma Center survivors were allowed to granulate and then closed with Vicryl mesh and split thickness skin grafting, this option is not recommended anymore due to improved laparostomy management. The performance of the decompressive laparotomy and the management of the open abdomen is described in the Appendix A of the SCALPEL Study Protocol - Best practice guideline for the decompressive laparotomy in the SCALPEL trial.

Follow up assessments:

GOS-E and EQ-5D will be evaluated at follow-up at 6 and 12 months in keeping with the IMPACT group recommendations. The investigators will use postal questionnaires, pre-paid envelopes, phone call reminders, structured phone call interviews and face-to-face interviews if necessary. The protocol does not allow members of the acute care team to participate in those interviews.

The questionnaires will be collected centrally, and two examiners will determine the outcome scores independently from each other.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. Traumatic Brain Injury with abnormal CT scan
3. Invasive ICP monitoring in place
4. ICP >25 mmHg for 1-12h after conventional therapies step I and step II (see Trial flow chart)

Exclusion Criteria:

1. Bilateral fixed and dilated pupil
2. Limitation of therapies by the team due to poor prognosis
3. Withdrawal of consent
4. Severe pre-existing physical or mental disability or co-morbidity which would lead to a poor outcome even if the patient made a full recovery from the head injury
5. Intracranial injury mandating craniotomy/craniectomy in itself
6. Intraabdominal injury mandating laparotomy in itself

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Functional outcome measured by the extended Glasgow Outcome Scale (GOS-E) | 12 months post-injury
  8 Good recovery Upper no current problems related to the brain injury that affect daily life; 7 Good recovery Lower minor problems that affect daily life; resumes >50% of the pre-injury level of social and leisure activities; 6 Moderate disability Upper reduced work capacity; resumes <50% of the pre-injury level of social and leisure activities; 5 Moderate disability Lower unable to work or only in sheltered workshop; 4 Sever disability Upper can be left alone > 8h during the day, but unable to travel and/or go shopping without assistance; 3 Sever disability Lower requires frequent help of someone to be around at home most of the time every day; 2 Persistent vegetative state unresponsive and speechless; 1 Death
  [higher scores mean better outcomes]

SECONDARY OUTCOMES:
Mortality | 30 days post-injury
Serious adverse events and surgical complications measured by the Clavien-Dindo Scale | 30 days post-injury
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition are also included.
  Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia
  Grade IV Life-threatening complication (including centralnervous complications)* requiring intensive care management
  * IVa single organ dysfunction (including dialysis)
  * IVb multi organ dysfunction Grade V Death of a patient
Frequency and severity of organ failure | 30 days post-injury
EQ-5D life quality | 6 and 12 months post-injury
  European Quality of Life Questionnaire [minimum 1, maximum 5, lower scores mean better outcomes]
GCS | 14 days post-injury
  Glasgow Coma Scale at discharge from intensive care [minimum 3, maximum 15; higher scores mean better outcomes]
Crossover-rate | 30 days post-injury
  Crossover-Rate: Participants who received an additional decompressive laparotomy after being randomly assigned to the decompressive craniectomy arm and Participants who received an additional decompressive craniectomy after being randomly assigned to the decompressive laparotomy arm.
Course of intracranial pressure | while in ICU for up to 14 days or until ICU discharge, whatever occurs first
  measured in mmHg
Intraabdominal pressure | while in ICU for up to 14 days or until ICU discharge, whatever occurs first
  measured in mmHg
Mean airway pressure | for up to 14 days or until ICU discharge, whatever occurs first
  measured in mbar
Hernia rate in the laparotomy group | 12 months post-injury
  rate of ventral incisional hernia post-laparotomy
Length of stay at the intensive care unit | up to 12 months
  measured in days
Length of stay at the neurosurgical unit | up to 12 months
  measured in days
Length of stay at the intensive care unit (ICU), neurosurgical unit, and rehabilitation unit | up to 12 months
  measured in days

CONTACTS AND LOCATIONS:
Locations (4):
- HIA Percy, Clamart, France
- Germany (3):
  - Bundeswehrzentralkrankenhaus Koblenz, Koblenz
  - Department of Neurosurgery - Klinikum rechts der Isar, Munich
  - Bundeswehrkrankenhaus Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolbel B, Novotny A, Willms A, Kehl V, Meyer B, Mauer UM, Krieg SM. Study protocol for a multicenter randomized controlled pilot study on decompressive laparotomy vs. decompressive craniectomy for intractable intracranial pressure after traumatic brain injury: The SCALPEL study. Brain Spine. 2023 Sep 26;3:102677. doi: 10.1016/j.bas.2023.102677. eCollection 2023. PMID 37822567